CLINICAL TRIAL: NCT06616402
Title: MOTU++ - Studio Clinico Protesi
Brief Title: Assessing the Usability and Reliability of the Prototype Prosthesis Devices
Acronym: MOTU++
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-PAI-02-23
Record Dates: First submitted 2024-09-02; First posted 2024-09-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-09

CONDITIONS: Amputation; Traumatic Amputations; Leg Amputation
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prosthetic group performs the entire protocol with the prosthesis prototype. (Other)
  Interventions: Device: prototype prosthetic group

INTERVENTIONS:
Device: prototype prosthetic group — These 3 sessions will commence only upon successful completion of the prosthesis safety and reliability tests conducted in the preceding sessions.
  For each module combination, a session will be conducted to assess motor performance through the acquisition of spatiotemporal parameters and energy efficiency parameters of gait. Motor performance will be evaluated using functional assessment tests and data will be recorded during the following activities:
  * parallel bar walking on flat ground
  * parallel bar walking on an inclined surface
  * treadmill walking with a safety harness
  * stair climbing/descending with a handrail
  * standing up and sitting down from a chair within parallel bars At the end of each session, satisfaction questionnaires (ad hoc questionnaire) will be completed. At the end of the experiment, a usability scale for the devices (ad hoc System Usability Scale) will be completed.
  Each session is expected to last approximately 2.5 hours.

SUMMARY:
The aim of the present study is to verify the functionalitỳ, the degree of safety and the reliability of devices composed of an intelligent socket that allows the detection of biosignals and provides vibrotactile feedback and a prosthesis with active knee and ankle joints and a sensorised foot, for people with trans-femoral or trans-tibial amputation, which allows the optimisation of the gait cycle by providing active assistance at the knee and ankle joints according to the specific movement made by the user. The prototype devices are innovative in that they make it possible to optimise the benefits generated by the presence of actuated joints by exploiting the biosignals detected to ensure optimal functionalitỳ in the performance of activities̀ of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* Lower limb amputation at the transfemoral or transtibial level;
* Functional medical classification: Level K3-K4 [25];
* Subjects wearing a prosthesis for at least 1 year (experienced wearers);
* Maximum body weight 100 kg.

Exclusion Criteria:

* Significant medical comorbidities: Presence of severe neurological disorders, cardiovascular diseases, uncontrolled diabetes/hypertension, or severe sensory deficits.
* Implanted cardiac devices: Individuals with implanted pacemakers or cardioverter-defibrillators.
* Cognitive impairment: Individuals with a Mini-Mental State Examination (MMSE) score less than 24, adjusted for age and education, indicating cognitive impairment that may compromise understanding of instructions and research participation.
* Severe depressive symptoms: Individuals with a Beck Depression Inventory-II (BDI-II) score less than 19, indicating clinically significant depression that may affect motivation and participation in the research.
* Severe anxiety symptoms: Individuals with a State-Trait Anxiety Inventory (STAI-Y) score less than 50, indicating clinically significant anxiety that may interfere with research participation.
* Inability or unwillingness to provide informed consent: Individuals who are unable to understand or provide informed consent to participate in the research, or who refuse to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Ad hoc check list for Adverse Event | baseline
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 1
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 2
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 3
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 4
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 5
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.
Ad hoc check list for Adverse Event | day 6
  questionnaire that evaluate the device feasibility of the prosthesis and description of any adverse events.

SECONDARY OUTCOMES:
Borg Scale | day 1
  0-10 numerical rating scale that evaluate of the subjective perception of efforts during walking.
Borg Scale | day 2
  0-10 numerical rating scale that evaluate of the subjective perception of efforts during walking.
Borg Scale | day 3
  0-10 numerical rating scale that evaluate of the subjective perception of efforts during walking.
Borg Scale | day 4
  0-10 numerical rating scale that evaluate of the subjective perception of efforts during walking.
Borg Scale | day 5
  0-10 numerical rating scale that evaluate of the subjective perception of efforts during walking.
10mwt - 10 meters walking test | baseline
  to evaluate walking capacity measured in seconds
10mwt - 10 meters walking test | day 4
  to evaluate walking capacity measured in seconds
6mwt - 6 minutes walking test | baseline
  to evaluate walking capacity measured in metres
System Usability Scale | day 6.
  a questionnaire made up of 10 questions whose answers are yes structured on a Likert scale with 0-100 that assesses the usability of the prosthesis.
TUG - Time Up and Go | baseline
  to assess lower limb capabilities in seconds
TUG - Time Up and Go | day 4
  to assess lower limb capabilities in seconds
SCT - Stair Climbing Test | baseline
  to assess the capabilities of climb 8 stairs in seconds
SCT - Stair Climbing Test | day 4
  to assess the capabilities of climb 8 stairs in seconds
6mwt - 6 minutes walking test | day 6
  to evaluate walking capacity measured in metres
FCT - Functional Reach Test | baseline
  to assess the balance in centimeters
Functional Reach Test | day 5
  to assess the balance in centimeters
Cost of Transport -COT | day 6
  To assess metabolic consumption

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No